CLINICAL TRIAL: NCT03849599
Title: A Phase 1b Study to Evaluate the Safety of PRV-300 Therapy in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Evaluate the Safety of PRV-300 in Adult Subjects With Moderately to Severely Active Ulcerative Colitis
Acronym: PULSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Provention Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRV-300-UC1b
Record Dates: First submitted 2019-02-17; First posted 2019-02-21 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2019-03

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group, multicenter study in adult subjects with moderately to severely active UC. Randomization will be stratified by Mayo score.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRV-300 (Experimental): Subjects in this arm will receive the study drug, PRV-300, via IV infusion, followed by an 8-week follow-up period.
  Interventions: Biological: PRV-300
- Placebo (Placebo Comparator): Subjects in this arm will receive placebo via IV infusion, followed by an 8-week follow-up period.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PRV-300 — Treatment
  Arms: PRV-300
Biological: Placebo — Control
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of PRV-300 for 12 weeks in subjects with active ulcerative colitis.

Subjects will receive either PRV-300 or placebo treatment. Each group will receive study drug over a total of 12 weeks, followed by an 8-week safety follow-up period.

DETAILED DESCRIPTION:
This is a Phase 1b, randomized, double-blind, placebo-controlled, parallel-group, multicenter study in adult subjects with moderately to severely active UC. Randomization will be stratified by Mayo score.

Subjects will receive either PRV-300 or placebo treatment. Each group will receive study drug over a total of 12 weeks, followed by an 8-week safety follow-up period. The total duration of the study will be 20 weeks, excluding the screening period.

The primary objective is to evaluate the safety and tolerability of PRV-300 for 12 weeks in subjects with active UC.

The secondary objectives are to evaluate the effect of PRV-300 for 12 weeks in subjects with active UC on:

* Pharmacodynamics: Changes in gene scores in colonic biopsies over the course of treatment.
* Pharmacokinetics: Peak (Cmax) and trough (Cmin) serum concentrations of PRV-300 in subjects with active UC.
* Immunogenicity: Immunogenicity of PRV-300 in subjects with active UC
* Endoscopic: Trends in endoscopic disease activity in subjects with active UC.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be a man or woman aged 18-75 years, inclusive.
2. Subject has a clinical diagnosis of UC at least 3 months before screening.
3. Subject has moderately to severely active UC, defined as a Mayo score of 6 to 12, inclusive, at screening.
4. Subject has a Mayo endoscopic subscore of ≥2 based on central read of the video sigmoidoscopy at screening.
5. Subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

1. Subject has severe extensive colitis as evidenced by any of the following:

   1. Current hospitalization for the treatment of UC.
   2. Investigator judgment that the subject is likely to require a colectomy within 12 weeks of baseline.
   3. Temperature ≥37.8 ºC (oral or tympanic) and a heart rate >90 bpm.
2. Subject has UC limited to <15 cm of the colon.
3. Subject has a diagnosis of CD or the presence or history of fistula or indeterminate colitis.
4. Presence of a gastrostomy, jejunostomy, ileostomy or colostomy.
5. Subject has had or is expected to have surgery for active gastrointestinal bleeding, peritonitis, intestinal obstruction, or intra-abdominal or pancreatic abscess requiring surgical drainage, or other conditions that may confound study evaluations from 2 months before screening through the end of this study.
6. Presence of symptomatic colonic or small bowel obstruction
7. History of colonic resection
8. History of colonic mucosal high-grade dysplasia
9. Subject has chronic or recurrent infectious disease
10. Subject has positive serology to human immunodeficiency virus (HIV) 1 or 2, hepatitis B virus (HBV) or hepatitis C virus (HCV) at screening.
11. Subject has any known malignancy or has a history of malignancy (with the exception of basal cell carcinoma; squamous cell carcinoma in situ of the skin; or cervical carcinoma in situ that has been treated with no evidence of recurrence; or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years before screening).
12. Subject has ever received PRV-300 (or CNTO 3157) or has known allergies, hypersensitivity, or intolerance to PRV-300 or its excipients; or known or suspected intolerance or hypersensitivity to any biologic medication or known allergies or clinically significant reactions to murine, chimeric, or human proteins, to monoclonal antibodies or antibody fragments; or a history of severe allergic reactions, angioedema, or anaphylaxis that might suggest risk for a reaction to a biologic agent.
13. Subject has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent adverse events (TEAEs), | 12 weeks
  Assessment of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Provention Bio, MD, Study Director — Provention Bio
Locations (3):
- Clinical Site, Tbilisi, Georgia
- Clinical Site, Chisinau, Moldova
- Clinical Site, Kapitanivka, Ukraine

IPD SHARING:
Plan to Share IPD: No